CLINICAL TRIAL: NCT02266550
Title: Investigation of Metabolism and Pharmacokinetics of [14C]-BIIL 284 BS After Administration of a Single Oral Dose of 25 mg [14C]-BIIL 284 BS in 6 Healthy Volunteers
Brief Title: Metabolism and Pharmacokinetics of [14C]-BIIL 284 BS in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 543.16
Record Dates: First submitted 2014-10-16; First posted 2014-10-17 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

INTERVENTIONS:
Drug: [14C] BILL 284 BS

SUMMARY:
The aims of this phase I study are to define the metabolism, excretion and pharmacokinetics of [14C]-BIIL 284 BS after administration of a single oral dose of 25 mg [14C]-BIIL 284 BS in 6 healthy volunteers. Tolerability was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, range from 30 to 55 years of age inclusive
* Body weight between 50 and 100 kg and within ± 20% of ideal body weight
* No clinically significant abnormal physical findings at the screening examination which would interfere with the objective of the study
* No clinically relevant abnormalities in the results of laboratory screening evaluation
* Normal ECG
* Normal Blood pressure (between 100 to 150 mmHg systolic and 50 to 90 mmHg diastolic) and heart rate (between 50 to 90 beats per minute)
* Able to communicate well with the investigator and to comply with the requirements of the entire study
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form
* Non-smokers

Exclusion Criteria:

* Medical examination or laboratory test results that are judged by the clinical investigator to differ significantly from normal clinical values
* Known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Current disease of the central nervous system (such as epilepsy) or with psychiatric disorders)
* Known history of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* Intake of any drugs which might influence the results of the trial during the week previous to the start of the study
* Administration of any investigational drug in the period 3 months before entry to the study (4 months if the previous drug was a new chemical entity)
* A need for any medication within the two weeks before dosing
* Existence of any surgical or medical condition which, in the judgement of the clinical investigator, might interfere with the absorption, distribution, metabolism or excretion of the drug (e.g. renal or hepatic impairments)
* Presence of clinically relevant history of allergy/hypersensitivity (including drug allergy)
* Blood loss or donation within the last 12 weeks (≥ 400 ml)
* Serious adverse reaction/hypersensitivity to any drug
* Objection by the subject's general practitioner to his/her patient's participation in the study
* Positive results for drug screening as listed in the protocol, positive results for hepatitis B surface antigen, Anti hepatitis B core antibodies, Anti hepatitis C virus antibodies and human immunodeficiency test, Glucose 6 - Phosphate Dehydrogenase
* Inability to communicate or co-operate with the investigator due to language problem, poor mental development or impaired cerebral function
* Administration of radiolabelled substance or exposure to significant radiation (e.g. serial X-ray, or CT scans, barium meal, etc) within the past 12 months
* History of recent drug abuse
* Volunteers who drink more than 4 units of alcohol per day and/or have been consuming alcohol during the 24 hours before dosing
* Participation in excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 1999-10; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Rates and routes of excretion of total radioactivity | up to 216 hours after drug administration
Concentration of [14C] radioactivity in blood | up to 216 hours after drug administration
Concentration of [14C] radioactivity in excreta (urine, faeces) | up to 216 hours after drug administration
Maximum concentration of the analytes in plasma (Cmax) | up to 216 hours after drug administration
Time to reach Cmax (tmax) | up to 216 hours after drug administration
Terminal half-life (t1/2) | up to 216 hours after drug administration
Mean residence time (MRT) | up to 216 hours after drug administration
Area under the drug concentration-time curve extrapolated from zero to infinity (AUC0-inf) | up to 216 hours after drug administration
Apparent clearance (CL/f) | up to 216 hours after drug administration
Volume of distribution (Vd/f) | up to 216 hours after drug administration
Nature of metabolites in plasma | up to 8 hours after drug administration
Nature of metabolites in urine | up to 48 hours after drug administration
Nature of metabolites in faeces | up to 48 hours after drug administration
Excretion balance on the basis of the [14C] radioactivity in urine and faeces | up to 216 hours after drug administration

SECONDARY OUTCOMES:
Number of subjects with clinically significant changes in laboratory parameters | up to 216 hours after drug administration
Number of subjects with clinically significant findings in physical examination | up to 216 hours after drug administration
Number of subjects with clinically significant changes in vital signs | up to 216 hours after drug administration
Number of subjects with clinically significant findings in 12-lead electrocardiogram | up to 216 hours after drug administration
Number of subjects with adverse events | up to 216 hours after drug administration